CLINICAL TRIAL: NCT04122768
Title: Enhancing Physical Activity in Patients After Lung Transplantation: Effectiveness and Feasibility of a Semi-automated Tele Coaching Program
Brief Title: Activity Coaching in Patients Post Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S62426
Record Dates: First submitted 2019-05-16; First posted 2019-10-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lung Transplantation
Keywords: physical activity; tele coaching; comorbidities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1 randomization. Patients who are active at baseline will not be randomized but will be followed up in a cohort study.
Who Masked: Participant
Masking Description: Patients in the control group will receive a sham version of the smartphone application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele coaching group (Experimental): Coaching with daily interaction with the coaching application, based on an adaptive physical activity goal
  Interventions: Behavioral: Multi-component physical activity tele coaching intervention
- Sham coaching group (Sham Comparator): Coaching with fixed physical activity goal and limited interaction with the smartphone application.
  Interventions: Behavioral: Light coaching intervention

INTERVENTIONS:
Behavioral: Multi-component physical activity tele coaching intervention — A.Education about the importance of PA. During a one-to-one interview with the coach motivation, self-efficacy, barriers, favorite activities and strategies to become more active are discussed.
  B. Step counter providing direct feedback.
  C.A smartphone with a project-tailored application. The application provides automated coaching by displaying an activity goal (number of steps) and feedback on a daily basis. The feedback comes with a graphical presentation. Patients' targets are automatically revised weekly. The aim is to progressively increase the PA during the 12 weeks period and maintain afterwards.
  D.Telephone contacts triggered in the case of non-compliance with wearing the step counter, failure to transmit data or failure to progress. Coaches are alerted by a note at the coaches' backend to take contact with the patient if needed.
  Arms: Tele coaching group
Behavioral: Light coaching intervention — A. Education about the importance of PA. During a one-to-one interview with the investigator, patients will receive a personal goal (expressed in steps/day), based on their individual exercise capacity.
  B.A step counter providing direct feedback.
  C.A smartphone with a project-tailored application. The application receives the step data of the patient and asks on a weekly basis about the patient's change in medication. The application does provide a graph showing the steps the patient took and presents a general activity plan including their personal goal (which stays the same throughout the entire intervention period).
  Arms: Sham coaching group

SUMMARY:
Lung transplantation is an ultimate, effective treatment option for selected patients with end stage lung disease, improving quality of life and extending survival. Because of the improved survival during the last decades, enhancing the long term condition after lung transplantation has now become a focus for disease management.

The co-presence of non-communicable diseases is common and poses new challenges to disease management. These comorbidities have been related to physical activity in the healthy population. As in other chronic respiratory disease, physical inactivity is a common feature of patients after LTX. Despite near normal lung function, exercise intolerance and physical inactivity persist up to years after the transplantation. Literature on effective interventions to increase physical activity are scarce in this population.

Therefore, the present project aims to test the effectiveness of a tele coaching program to enhance physical activity and to analyze the association between physical activity and long-term health benefits in this population at risk. These research questions will be answered based on a randomized controlled trial. Patients that are active at baseline will be followed up in a cohort study.

DETAILED DESCRIPTION:
The aims of the present study are:

1) primary objective: To test the effectiveness of adding a semi-automated tele coaching intervention to enhance physical activity in patients after a first double lung transplantation, assessed at 12 weeks.

2) Secondary objectives:

1. To test the long term effect of a semi-automated tele coaching intervention on physical activity, assessed at 52 weeks.
2. To analyze the association between baseline physical activity, the change in physical activity and long term health benefits in this population at risk
3. To relate the day-by-day pattern of physical activity to changes in the health status of patients.
4. To investigate the patient's experience with the delivered intervention.

Therefore, the study will include stable patients at least 6 months and maximum 4 years after a first double lung transplantation. Based on a 1 week physical activity assessment, patients will be classified as active (mean steps >7500 steps) or inactive (mean steps < 7500). Inactive patients will be entered in a randomized controlled trial, using block randomization. Active patients will be followed for 1 year in a cohort study.

The study consists of a total of 3 (active patients) or 4 (inactive patients) clinical visits:

* Visit 1 screening visit (all patients)
* Visit 2: randomisation visit, scheduled 1-2 weeks after visit 1 (all patients)
* Visit 3: short term follow up, scheduled 12 weeks after visit 2. T(only in patients who have been randomized)
* Visit 4: long term follow up, scheduled 52 weeks after visit 2. (all patients)

Active patients will be measured again 52 weeks after visit 2. They will not receive any intervention during the 1 year follow up. Patients who enter the randomized controlled trial will either receive

* A mulitcomponent tele coaching intervention that consists of 1) education about the importance of physical activity and a one-to-one interview with the coach discussing motivation and barriers to be active, 2) a step counter providing direct feedback, 3) application installed on a smartphone providing an adaptive goal and daily and weekly feedback and 4) contact with the coach if the patient is not compliant with the intervention, not increasing physical activity or when the patient reports a change in medication. The patient is asked to have a daily interaction with the smartphone application.
* A sham intervention that consist of 1) education about the importance of physical activity and a personal (fixed) goal expressed in terms of steps. The patient is asked to try to reach this goal, 2) a step counter providing direct feedback, 3) application installed on a smartphone only displaying a graph with the activity of the present week and the personal (fixed) goal, 4) contact with the coach if the patient reports a change in medication. The patient is asked to have at least a weekly interaction with the application.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients at least 6 months and maximum 4 years after the first double lung transplantation
2. Older than 30 years
3. Understand and able to work with the smartphone application, as judged by the investigator

Exclusion Criteria:

1. Having a diagnosis of Cystic Fibrosis
2. Musculoskeletal problems not allowing a normal gait pattern
3. Receiving a multi-organ transplantation or previously undergoing a solid-organ or bone marrow transplantation
4. Chronic rejection of the allograft before inclusion
5. Having a life expectancy <1year

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Daily number of steps at 12 weeks (short term effect) | 12 weeks
  Change in daily mean step count 12 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.

SECONDARY OUTCOMES:
Proportion of responders | 12 weeks and 52 weeks
  Proportion of patients showing an increase of at least 1000 steps. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Daily number of steps at 52 weeks (long term effect) | 52 weeks
  Change in daily mean step count 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Exercise capacity | 12 weeks and 52 weeks
  Change in six-minutes walk distance 12 and 52 weeks post randomization in the intervention group as compared to the control group. The six-minute walking test will be performed with standardized encouragement to assess patients' functional exercise capacity. The best of two measurements will be used.
Quadriceps force | 12 weeks and 52 weeks
  Change in isometric quadriceps force 12 and 52 weeks post randomization in the intervention group as compared to the control group. The quadriceps isometric strength will be evaluated by a maximal voluntary contraction using the Biodex, a computerized dynamometer. Patients will be seated with a 90° hip and 60° knee flexion. The best of 3 measurements will be taken into analysis as the maximal force capacity of the lower limb.
Health related quality of life | 12 weeks and 52 weeks
  Change in quality of life 12 and 52 weeks post randomization in the intervention group as compared to the control group. Health related quality of life will be measured by the extensively validated generic HRQoL questionnaire, the SF-36. This questionnaire includes two main scores with a physical component and an emotional component scale and eight subscales.
Symptoms of anxiety and depression | 12 weeks and 52 weeks
  Change in symptoms of anxiety and depression 12 and 52 weeks post randomization in the intervention group as compared to the control group. Symptoms of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADs). The HADs is a generic screening measure of symptoms of anxiety and depression. The HADS is a 14 item measure comprising 7 anxiety items and 7 depression items from which separate anxiety and depression sub-scale scores are calculated.
Symptoms of fatigue | 12 weeks and 52 weeks
  Change in symptoms of fatigue 12 and 52 weeks post randomization in the intervention group as compared to the control group. Fatigue will assessed using the subscale fatigue of the Checklist Individual Strength (CIS). The subscale consists of 8 items. Each item is scored on a 7-point scale. The total score ranging from 8 to 56 is calculated. Significant fatigue is defined as a score of 35 or higher on the CIS fatigue.
Time spent in at least moderate intense activity | 12 weeks and 52 weeks
  Change in daily time spent in at least moderate intense activity 12 and 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Mean walking time per day | 12 weeks and 52 weeks
  Change in mean daily walking time 12 and 52 weeks post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in in chronic respiratory disease. Data obtained on days with more than 8 hours of wearing time will be used for further analysis.
Metabolic syndrome | 52 weeks
  Prevalence of abdominal obesity, hyperlipidemia, hypertension and diabetes (and combined in the metabolic syndrome). Abdominal obesity will be assessed by waist and hip circumference, hypertension will be assessed by 2 tests of blood pressure with at least 5 minutes interval, hyperlipidemia and diabetes will be assessed based on a fasted blood sample.
Lipid profile | 52 weeks
  Serum lipid profile (total cholesterol, triglyceride, HDL and LDL) based on a fasted blood sample
blood pressure | 52 weeks
  Blood pressure will be assessed twice with at least 5 minutes interval
ankle brachial index | 52 weeks
  Peripheral vascular disease will be assessed by the ankle brachial index as the ratio between the blood pressure in the arms and the blood pressure in the lower legs.
Body mass index | 52 weeks
  Calculated as the ratio between weight and height (squared)
Body composition | 52 weeks
  Fat free and fat mass based on DEXA scan
Waist and hip circumference | 52 weeks
HOMA IR | 52 weeks
  Calculated based on glucose and insuline levels measured during a fasted blood sample
HbA1c | 52 weeks
  HbA1c based on fasted blood sample
bone mineral density | 52 weeks
  Bone mineral density measured by DEXA scan
Systemic inflammation | 52 weeks
  CRP based on a blood sample.
vitamin D level | 52 weeks
  vitamin D levels based on a blood sample.
Cardiopulmonary exercise test (only in patients 6-9 months post transplantation) | 52 weeks
  Maximal exercise capacity will be assessed by a maximal incremental cycling test (Ergometrics 900, Ergoline, Bitz, Germany). After a 2-min resting period and 3 minutes of unloaded cycling, the patients will start at 20 W and cycle until symptom limitation at an incremental workload of 10 W/min. Oxygen consumption, carbon dioxide output and ventilation will be measured breath by breath (Vmax series, SensorMedics, Anaheim, CA). Heart rate and oxygen saturation will be registered continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Troosters, Prof, Principal Investigator — KU Leuven; Heleen Demeyer, Dr, Principal Investigator — KU Leuven; Wim Janssens, Prof, Principal Investigator — KU Leuven; Robin Vos, Prof, Principal Investigator — KU Leuven; Daniel Langer, Prof, Principal Investigator — KU Leuven; Geert Verleden, Prof, Principal Investigator — KU Leuven
Locations (1):
- KULeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Breuls S, Blondeel A, Wuyts M, Verleden GM, Vos R, Janssens W, Troosters T, Demeyer H. 1-year physical activity coaching programme in lung transplant recipients: an RCT. Thorax. 2025 Sep 15;80(10):711-719. doi: 10.1136/thorax-2024-222896. PMID 40447328